CLINICAL TRIAL: NCT03934437
Title: Leveraging mHealth and Peers to Engage African-Americans and Latinxs in HIV Care (LEAN)
Brief Title: Leveraging mHealth and Peers to Engage African- Americans and Latinxs in HIV Care (LEAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00195120; 11244 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mLTCR (Experimental): The mLTCR intervention consists of two smartphone applications (app), one for patients and one for patient supporters, to help facilitate communication.
  Interventions: Behavioral: mLTCR
- LTC (Active Comparator): Existing linkage to care and retention (LTCR) services which are standard-of-care
  Interventions: Behavioral: LTCR

INTERVENTIONS:
Behavioral: mLTCR — mHealth-enhanced Linkage to Care and Retention
  Arms: mLTCR
Behavioral: LTCR — Linkage and Retention Services (Standard-of-Care)
  Arms: LTC

SUMMARY:
This is a pragmatic randomized controlled study comparing existing linkage to care and retention (LTCR) services to an mHealth-enhanced linkage to care and retention (mLTCR) protocol.

DETAILED DESCRIPTION:
Baltimore's HIV prevalence rate (586/100,000) is among the top 5 in metropolitan areas in the US, and disparities are profound. African Americans have an HIV prevalence that is 5 times higher than among whites, and account for 78% of all HIV cases. Latinxs also have a higher prevalence of HIV than whites and are at the highest risk for late HIV diagnosis among all racial/ethnic groups. In addition, HIV viral load suppression, which is the best predictor of long-term survival among HIV-infected patients, is substantially lower among minority populations in Baltimore.

The overall goal of this proposal is to evaluate whether mHealth-enhanced Linkage to Care and Retention (mLTCR) can improve HIV outcomes among HIV-infected African Americans and Latinos compared to standard Linkage to Care and Retention (LTCR) programs. The mHealth-enhancement consists of two smartphone applications (app), one for patients and one for patient supporters (e.g. linkage officers, patient navigators, nurses, etc.), to help facilitate communication. Communication will focus on issues related to HIV care (e.g. appointment scheduling, transportation), as well as patient-directed requests. Using HIV surveillance data (e.g. unsuppressed HIV viral load), patient supporters will be automatically alerted if a patient has a high viral load and prompted to contact the patient. In addition to appointment reminders, patients will receive positive reinforcement behavioral text messages.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Ability to provide consent
* Identified by BCHD Linkage protocol to be a new HIV diagnosis or HIV-infected and "out of care"
* Identified by participating clinics as needing patient support services

Exclusion Criteria:

* Not able to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen W Page, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Baltimore City Health Department, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for data sharing should be made to the PI.
Supporting Information: Study Protocol
Time Frame: Within 1 year after study recruitment has begun.
Access Criteria: All reasonable requests will be considered.

REFERENCES:
- [Derived] Jones J, McKenzie-White J, Saxton R, Grieb SM, Nonyane B, Graham C, Cano A, Johnson S, Childs L, Greenbaum A, Flynn C, Pearlowitz M, Celano S, Chang LW, Page KR. Leveraging mHealth and Patient Supporters for African Americans' and Latinxs' Engagement in HIV Care (LEAN): Protocol for a Randomized, Controlled, Effectiveness-Implementation Trial. JMIR Res Protoc. 2023 Feb 14;12:e42691. doi: 10.2196/42691. PMID 36787165

RESULTS

PARTICIPANT FLOW:
Groups:
- LTCR: Existing linkage to care and retention (LTCR) services which are standard-of-care
  LTCR: Linkage and Retention Services (Standard-of-Care)
Period: Overall Study
Arm/Group | mLTCR | LTCR
Started | 225 | 226
Completed | 223 | 225
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: 3 participants withdrew.
Groups:
- Total: Total of all reporting groups
Arm/Group | mLTCR | LTCR | Total
Number analyzed (Participants) | 223 | 225 | 448
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 210 | 207 | 417
  >=65 years | 13 | 18 | 31
Age, Continuous [Mean (Full Range); unit: years] | 45.1 [21 to 70] | 45.0 [20 to 78] | 45.1 [20 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 73 | 160
  Male | 136 | 152 | 288
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 6 | 8
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 173 | 172 | 345
  White | 20 | 17 | 37
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 22 | 25 | 47
Region of Enrollment [Number; unit: participants]
  United States | 223 | 225 | 448
HIV Viral Load Suppression (Copies/cc) [Count of Participants; unit: Participants] — Viral Suppression defined as a viral load < 200 copies/cc
  Participants
    Undetectable (<200 copies/cc, well controlled) | 112 | 128 | 240
    Detectable (>=200 copies/cc, poorly controlled) | 93 | 82 | 175
    No VL (presumed poorly controlled) | 18 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Participants With HIV Viral Load Suppression (Copies/cc)
Description: Viral Suppression defined as a viral load < 200 copies/cc
Time Frame: 12 months
Population: Two participants withdrew from mLTCR; one participant withdrew from LTCR.
Measure: Count of Participants; unit: Participants
Arm/Group | mLTCR | LTCR
Number analyzed (Participants) | 223 | 225
Participants
  Undetectable (<200 copies/cc, well controlled) | 114 | 128
  Detectable (>=200 copies/cc, poorly controlled) | 38 | 32
  No VL (presumed poorly controlled) | 71 | 65

2. Secondary Outcome: Participants Retained in Care
Description: Retained in care based upon viral load, CD4, OR clinic visit reported in enhanced HIV/AIDS Reporting System (eHARS)
Time Frame: 12 months
Population: Two participants withdrew from mLTCR; one participant withdrew from LTCR.
Measure: Count of Participants; unit: Participants
Arm/Group | mLTCR | LTCR
Number analyzed (Participants) | 223 | 225
Participants | 152 | 160

ADVERSE EVENTS:
Time Frame: Up to 12 months
Groups:
- Linkage to Care: Existing linkage to care and retention (LTCR) services which are standard-of-care
  LTCR: Linkage and Retention Services (Standard-of-Care)
Arm/Group | mLTCR | Linkage to Care
All-Cause Mortality (participants affected / at risk) | 9/225 | 11/226
Serious Adverse Events (participants affected / at risk) | 0/225 | 0/226
Other Adverse Events (participants affected / at risk) | 0/225 | 0/226

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03934437/Prot_SAP_000.pdf